CLINICAL TRIAL: NCT00598507
Title: Phase II Trial Of ZK-EPO (ZK 219477) (Sagopilone) In Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14965; ZK219477 (Other: Berlex); 108.0701 (Other: Bayer Corporation)
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-08

CONDITIONS: Melanoma
Keywords: ZK-EPO; ZK219477; EpothiloneZK
MeSH Terms: conditions — Melanoma | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy - ZK-EPO (Experimental): ZK-EPO (ZK 219477) (Sagopilone), 16 mg/m^2, was administered intravenously over 3-hours every 21 days until progression or unacceptable toxicity.
  Interventions: Drug: ZK-EPO

INTERVENTIONS:
Drug: ZK-EPO — Participants were treated with 16 mg/m^2 of ZK-EPO (EpothiloneZK) (Sagopilone) administered as a single 3 hour intravenous infusion every 21 days. Prior to each treatment, participants were premedicated with either granisetron or ondansetron and additional anti-emetics if needed. Chemotherapy was continued until disease progression, withdrawal of consent, or for unacceptable treatment-associated toxicity.
  Other Names: EpothiloneZK; ZK 219477; Sagopilone

SUMMARY:
The purpose of this study is to find out how effective an investigational drug named ZK-Epo is against melanoma. Although ZK-Epo has been studied in the treatment of cancer, it is not approved for use in treating melanoma. This research is being done because currently there are only a limited number of treatment options for patients who have melanoma that has spread to distant organs.

We expect each patient to be in this study for at least 2 cycles. One cycle lasts for 21 days. If their tumor does not grow after 2 cycles and they do not have any major side-effects, they may receive up to 6 cycles of ZK-Epo.

If after they have received 6 cycles of ZK-Epo and their doctor determines that the tumor is continuing to shrink, they will continue treatment with ZK-Epo. The number of treatments the patient receives after 6 cycles will depend upon when their doctor feels there has been maximum tumor response (tumor shrinkage). Two treatments will be given beyond what their doctor considers the point of maximum shrinkage. We estimate that they will spend anywhere from 1 1/2 months to 5 months taking part in this study.

DETAILED DESCRIPTION:
Each Cycle is a 21 day period. On the first day of each cycle each patient will receive the study drug, ZK-Epo, through an IV infusion over a 3 hour period. Patients will receive the study drug only once every 21 day period.

At the start of each cycle patients will have the following tests:

* Patients will be asked questions about their medical history and health and undergo a complete physical exam.
* Blood tests will be done to check blood cell count and organ functions (about 1 tablespoon of blood will be taken).
* Performance status tests (will determine patient's ability to perform everyday functions).
* A nurse or doctor will ask patients how they are feeling and about any side effects that patients may be having.
* Pre Study Visit: Blood test called lactate dehydrogenase (LDH) to check organ function. Prothrombin time (PT) and an a partial thromboplastin time (PTT) to see if the patient's blood clots normally. Electrocardiogram (EKG) (to measure the electrical function of patient's heart). Pregnancy Test (IF APPLICABLE a woman of child bearing age). Optional Tumor Biopsy (If indicated by patient's physician).
* Cycle 1, Day 1: Pharmacokinetics: special blood tests to measure the drug levels, LDH
* Cycle 1, Day 2 & 8: Pharmacokinetics
* Cycle 1, Day 15: EKG
* Cycle 2, DAY 1: LDH
* Cycle 3, DAY 1: LDH, PT & activated partial thromboplastin time (aPTT)
* Cycle 4, 5, & 6, and all subsequent cycles, Day 1: LDH

During the first cycle only patients will also need to come for a study visit on day 8 and 15. During these two visits, blood tests will be done again to check blood cell count and organ functions. Patients will also be asked how they are feeling and about any side effects that they may be having.

Computed tomography (CT) scans or a magnetic resonance imaging (MRI) will be done after every 2 cycles that each patient completes on the study. These will be done to help the doctor re-evaluate each patient's disease.

Patients may have some additional blood tests done if they are among the first 10 patients taking part in this study. In this case they will have 9 samples of blood (each about a teaspoonful) drawn from them at specifically timed intervals (at 30 minutes before the start and at 30 minutes, 2 hour 55 minutes, 3 hour 10 minutes, 3 hour 30 minutes, 5 hour, 8 hour, 27 hour (+/- 1 hour) and 168 hour (+/- 4 hours) after the start of the ZK-Epo infusion) so that we can better understand the level of this drug in the body and its metabolism in people.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Malignant Melanoma.
* Unresectable Stage III or Stage IV disease.
* At least 1 measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Adequate function of major organs and systems as measured by the following criteria:

Bone Marrow:

* Hemoglobin ≥ 10 g/dL
* White blood count (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin within 1.5 times normal limit
* aspartate transaminase (AST)/Alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN)

Renal:

* Creatinine ≤ 2 mg/dL

Cardiovascular:

* No New York Heart Association (NYHA) class III or IV Congestive heart failure
* No unstable angina pectoris
* No arrhythmia needing continuous treatment

Nervous system:

* No Grade ≥ 2 peripheral neuropathy

Exclusion Criteria:

* More than 2 previous chemotherapy regimens.
* Any prior treatment with Epothilones, Epothilone analogues, taxanes, or vinca alkaloids.
* Any progressive central nervous system (CNS) metastatic disease. Patients with CNS metastases may be allowed if stable for 8 weeks or more and patient is neurologically intact and off of steroids. The stability must be documented by MRI/CT over a period of 8 weeks or greater.
* Any radiotherapy, chemotherapy, or immunotherapy within 3 weeks prior to first dose of ZK-Epo. If patients were previously on temozolomide with extended dose schedule, they must be off 1 week prior to the first dose of ZK-Epo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeConti, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual began in May 2007 at Moffitt Cancer Center and was completed in October 2008.
Period: Overall Study
Arm/Group | Chemotherapy - ZK-EPO
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants treated with at least one dose of sagopilone.
Arm/Group | Chemotherapy - ZK-EPO
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 23
Age Continuous [Median (Standard Deviation); unit: years] | 68.7 (1.7) [37 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Objective tumor response according to Response Evaluation Criteria In Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 5 years
Population: All participants
Measure: Number; unit: participants
Arm/Group | Chemotherapy - ZK-EPO
Number analyzed (Participants) | 35
participants
  Confirmed Complete Response | 1
  Confirmed Partial Response | 2
  Unconfirmed Partial Response | 1
  Stable Disease for at Least 12 Weeks | 8

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS: the duration of time from start of treatment to time of progression or death, whichever occurs first. Progressive Disease (PD)according to modified Response Evaluation Criteria in Solid Tumors (RECIST) Criteria: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 5 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy - ZK-EPO
Number analyzed (Participants) | 35
weeks | 7.5 [6.4 to 8.7]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Median OS: the time (expressed in months or years) when half the patients are expected to be alive.
Time Frame: Up to 5 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy - ZK-EPO
Number analyzed (Participants) | 35
weeks | 31 [14.9 to 47.1]

4. Secondary Outcome: Occurrence of Attributable Serious Adverse Events (SAEs)
Description: Number of participants with Grade 3 or higher adverse events, attributable to treatment with sagopilone.
Time Frame: Up to 5 years
Population: All participants
Measure: Number; unit: participants
Arm/Group | Chemotherapy - ZK-EPO
Number analyzed (Participants) | 35
participants | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Participants treated with at least one dose of sagopilone.
Arm/Group | Chemotherapy - ZK-EPO
Serious Adverse Events (participants affected / at risk) | 5/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy - ZK-EPO (N=35)
Confusion (General disorders) | 1
Creatinine - high (Metabolism and nutrition disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Fever in the absence of neutropenia (General disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Pulmonary hypertension (Cardiac disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Syncope (fainting) (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy - ZK-EPO (N=35)
Neuropathy: sensory (Nervous system disorders) | 19
Neuropathy: motor (Nervous system disorders) | 8
Confusion (General disorders) | 2
Hemoglobin - low (Blood and lymphatic system disorders) | 11
Leukocytes (total WBC) - low (Blood and lymphatic system disorders) | 8
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 5
Platelets - low (Blood and lymphatic system disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13
Fever (in the absence of neutropenia) (General disorders) | 3
Constitutional Symptoms - Other (General disorders) | 2
Pain - Extremity-limb (General disorders) | 7
Pain - Joint (General disorders) | 7
Pain - Muscle (General disorders) | 5
Pain - Back (General disorders) | 3
Pain - Bone (General disorders) | 2
Pain - Head/headache (General disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) - high (Metabolism and nutrition disorders) | 2
AST, SGOT(serum glutamic oxaloacetic transaminase) - high (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Anorexia (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Hypotension (Cardiac disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Lymphatic (Infections and infestations) | 2
Edema: limb (Blood and lymphatic system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes